CLINICAL TRIAL: NCT02071758
Title: A Phase 1, Open-Label Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of the LEISH-F3 + SLA-SE Vaccine Compared to LEISH-F3 + GLA-SE Vaccine in Healthy Adult Subjects
Brief Title: Phase 1 LEISH-F3 + SLA-SE Vaccine Trial in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDRI-LVVPX-117
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Visceral Leishmaniasis
Keywords: Leishmaniasis; Visceral leishmaniasis; Vaccine; Adjuvant; GLA; SLA
MeSH Terms: conditions — Leishmaniasis, Visceral; Leishmaniasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 20 mcg LEISH-F3 + 5 mcg SLA-SE Vaccine (Experimental): Three intramuscular injections of LEISH-F3 + SLA-SE at Days 0, 28, and 56. High dose of antigen and low dose of SLA-SE adjuvant.
  Interventions: Biological: LEISH-F3 + SLA-SE
- 20 mcg LEISH-F3 + 10 mcg GLA-SE Vaccine (Experimental): Three intramuscular injections of LEISH-F3 + GLA-SE at Days 0, 28, and 56. High dose of antigen and high dose of GLA-SE adjuvant.
  Interventions: Biological: LEISH-F3 + GLA-SE
- 5 mcg LEISH-F3 + 10 mcg GLA-SE Vaccine (Experimental): Three intramuscular injections of LEISH-F3 + GLA-SE at Days 0, 28, and 56. Low dose of antigen and high dose of GLA-SE adjuvant.
  Interventions: Biological: LEISH-F3 + GLA-SE
- 20 mcg LEISH-F3 + 10 mcg SLA-SE Vaccine (Experimental): Three intramuscular injections of LEISH-F3 + SLA-SE at Days 0, 28, and 56. High dose of antigen and high dose of SLA-SE adjuvant.
  Interventions: Biological: LEISH-F3 + SLA-SE

INTERVENTIONS:
Biological: LEISH-F3 + SLA-SE
  Arms: 20 mcg LEISH-F3 + 10 mcg SLA-SE Vaccine; 20 mcg LEISH-F3 + 5 mcg SLA-SE Vaccine
Biological: LEISH-F3 + GLA-SE
  Arms: 20 mcg LEISH-F3 + 10 mcg GLA-SE Vaccine; 5 mcg LEISH-F3 + 10 mcg GLA-SE Vaccine

SUMMARY:
The purpose of this study is to compare the safety, tolerability, and immunogenicity in healthy adult subjects of an investigational vaccine being developed for the prevention of visceral leishmaniasis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 49 years of age.
* Must be in good general health as confirmed by a medical history and physical exam.
* Female subjects must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of each study vaccination, must not be breast-feeding, and are required to use one of the following methods of contraception during the first 3 months of the study: hormonal (e.g., oral, transdermal, intravaginal, implant, or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD) or system (IUS); vasectomized partner (6 months minimum); abstinence; or bilateral tubal ligation (if no conception post-procedure). These precautions are necessary due to unknown effects that LEISH-F3 + SLA-SE or LEISH-F3 + GLA-SE might cause in a fetus or newborn infant.
* The following screening laboratory values must be within the normal ranges or not clinically significant as determined by the PI and Medical Monitor (MM): sodium, potassium, BUN, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, fasting glucose, total WBC count, hemoglobin, and platelet count.
* The following serology tests must be negative: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
* Negative urine test for recreational drugs and alcohol per Clinical Research Unit standards.
* Urinalysis not clinically significant as determined by the study clinician.
* Must be capable of completing a study memory aid in English.
* Must give informed consent, be able and willing to make all evaluation visits, be reachable by telephone or personal contact by the study site personnel, and have a permanent address.

Exclusion Criteria:

* History of possible infection with Leishmania or previous exposure to Leishmania vaccines or experimental products containing SLA or GLA.
* Veterans who served in the military in the Middle East (Iran, Iraq), Afghanistan, or any other areas endemic to Leishmania.
* Travelers to, or immigrants from, areas endemic to Leishmania.
* Participation in another experimental protocol or receipt of any investigational products within the past 3 months.
* Treatment with immunosuppressive drugs (e.g., oral or injected steroids, such as prednisone; high dose inhaled steroids) or cytotoxic therapies (e.g., chemotherapy drugs or radiation) within the past 6 months.
* Received a blood transfusion within the past 3 months.
* Donated blood products (platelets, whole blood, plasma, etc.) within past one month.
* Received any vaccine within past 1 month and no planned immunizations while on study with the exception of seasonal influenza vaccine which should not be given between Day 0-84 or Day 138-168 due to 30-day washout period prior to immunology blood draws.
* History of autoimmune disease or other causes of immunosuppressive states.
* History or evidence of any acute or chronic illness (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic, or renal disorders, controlled hypertension), or use of medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Rash, tattoos, or any other dermatological condition that could adversely affect the vaccine injection site or interfere with its evaluation.
* BMI, that in the opinion of the Investigator, poses a health risk.
* Hypertension (systolic >150 or diastolic >95).
* History of significant psychiatric illness with current use of medication.
* Known or suspected alcohol or drug abuse within the past 6 months.
* Chronic smoker (> 20 pack years).
* Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines, eggs, or unknown allergens.
* Subjects who are unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 421 days
  Solicited and unsolicited adverse events will be recorded for 28 days following each study injection; serious adverse events and adverse events of special interest will be recorded for the duration of the study.

SECONDARY OUTCOMES:
Immunogenicity | Days 0, 7, 35, 63, 84, and 168
  Immunogenicity will be evaluated by measuring humoral and cellular responses to LEISH-F3 + SLA-SE or LEISH-F3 + GLA-SE at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Marie Beckmann, PhD, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Covance, Inc., Daytona Beach, Florida, United States